CLINICAL TRIAL: NCT05552729
Title: Effect of Different Doses of Vitamin D on Cancer-related Cognitive Impairment in Patients With Gastrointestinal Tumors: a Randomized Controlled Study
Brief Title: Effects of Different Doses of Vitamin D on Cancer-related Cognitive Impairment in Patients With Gastrointestinal Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yangzhou University (Other)
Collaborators: Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Principal Investigator, Wang Daorong, Professor, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yangzhou University
Record Dates: First submitted 2022-09-03; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Neoplasms; Cognitive Impairment
Keywords: Gastrointestinal Neoplasms; Cognitive Impairment; Vitamin D
MeSH Terms: conditions — Gastrointestinal Neoplasms; Cognitive Dysfunction | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Active Comparator): A 2000IU vitamin D3 supplement was started the next day after surgery.
  Interventions: Drug: Vitamin D
- Low dose group (Active Comparator): A 400IU vitamin D3 supplement was started the next day after surgery.
  Interventions: Drug: Vitamin D
- The control group. (No Intervention): No vitamin D3 supplement was started the next day after surgery.

INTERVENTIONS:
Drug: Vitamin D — The patients were given vitamin D supplementation 48 hours after surgery, and the two groups were given different doses of vitamin D supplementation until the postoperative discharge criteria were met. To scientifically evaluate the application effect of early postoperative vitamin D intervention in the improvement of perioperative cognitive function in patients with gastrointestinal tumors.
  Other Names: Different doses of vitamin D
  Arms: High dose group; Low dose group

SUMMARY:
To explore the effect of different doses of vitamin D drugs on gastrointestinal cancer cancer-related cognitive impairment, so as to provide reference and basis for the clinical use of our cognitive function surgery nursing plan for patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
To determine the incidence of postoperative cognitive dysfunction in patients with gastrointestinal tumors to determine the influencing factors of postoperative cognitive dysfunction in patients with gastrointestinal tumors. The characteristics of perioperative cancer-related cognitive impairment in patients with gastrointestinal tumors were analyzed by monitoring preoperative and postoperative FACT-COG cognitive scale connection test (Hua-Shan-version auditory word learning test) DSST digit symbol test gaffes detection task and hematology indexes, such as observation and analysis of the interference pattern of supplement vitamin D preparation postoperative hospital stay in patients with gastrointestinal tumor short-term cognitive impairment related to cancer, in order to reduce the incidence of complications and hospitalization days, improve cognitive function in patients with gastrointestinal tumor surgery, and improve the quality of nursing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastrointestinal tumors diagnosed by gastroscopy and histology and their family members
* Elective surgery
* Education level in primary school or above
* Be able to fill in the questionnaire alone or under the guidance of the researcher
* Informed consent and voluntary participation in this study

Exclusion Criteria:

* Patients with cognitive impairment (illiteracy less than 17 points, primary school less than 20 points, secondary school or above less than 24 points) or previous history of cognitive impairment, dementia and delirium confirmed by MMSE examination before surgery
* Patients with life-threatening acute and chronic diseases
* Patients with eye or ear diseases leading to rapid loss of hearing or vision without AIDS
* Patients who have taken drugs related to improving cognitive function or drugs for psychiatric disorders
* Patients who cannot take care of themselves or are physically disabled and unable to perform neurological function tests
* Intraoperative hypoxemia (blood oxygen saturation < 94％) more than 10 minutes
* Patients who quit or died due to non-cooperation or emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-09-22 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Eight days after the surgery
  Fact-cog Cognitive Scale.The higher the score, the better the cognition.

SECONDARY OUTCOMES:
Sleep | Eight days after the surgery
  Pittsburgh sleep quality index.The overall score ranges from 0 to 21, with a score of 0 to 5 indicating good sleep quality,6 to 10 indicating fair sleep quality,11 to 15 indicating fair sleep quality, and 16 to 21 indicating very poor sleep quality.
Cancer related fatigue | Eight days after the surgery
  Cancer Fatigue Scale. The total score ranges from 0 to 15, and 4 is considered frailty.
Asthenia | Eight days after the surgery
  Groningen Frailty Indicator. The total score ranges from 0 to 15, and 4 is considered frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Daorong Wang, Professor, Study Director — Yangzhou University
Locations (1):
- Daorong Wang, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No